CLINICAL TRIAL: NCT07355985
Title: Multi-omics Analysis of Prostate Derived Extracellular Vesicles: an Observational Retrospective Study for Prostate Cancer Diagnosis and Monitoring
Acronym: EXOMAP
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Alberto Briganti, Full Professor, IRCCS San Raffaele
Other Study IDs: EXOMAP
Record Dates: First submitted 2025-12-10; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer Adenocarcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prostate cancer (PCa) is the most commonly diagnosed malignancy in men and a leading cause of cancer-related mortality worldwide. Over 1.4 million new cases of prostate cancer are estimated to occur worldwide each year, with more than 375,000 related deaths. High-risk PCa poses significant challenges due to the aggressive nature of the disease and the ability to create an immunosuppressive tumor microenvironment (TME), thereby hampering the effectiveness of existing therapies. Despite advances in diagnostics and treatment, the mechanisms driving immune evasion and tumor progression in high-risk PCa remain poorly understood. These considerations underscore the urgent need for innovative strategies to address these challenges and improve patient outcomes.

Extracellular vesicles (EVs) have emerged as critical players in cancer biology. EVs carry molecular cargo, including proteins, RNA, lipids, and metabolites, enabling mediation of intercellular communication and influence on cancer progression. Tumor-derived EVs (TDEVs) are particularly implicated in promoting tumor growth, reprogramming the TME, and suppressing antitumor immune responses. Owing to the intrinsic ability to mediate intercellular communication and transport biomolecules to distant sites, EVs represent key contributors to cancer pathogenesis.

A previous study demonstrated, through comprehensive metabolomics profiling, a combination of small molecules extracted from expressed prostatic secretion (EPS)-urine, integrated with clinical parameters, that could effectively identify and stratify PCa patients, highlighting the potential of this biofluid in PCa diagnostics. EPS-urine represents a unique biofluid enriched with EVs secreted directly by prostate tissue, offering a valuable source for the study of prostate-specific EVs. Based on this evidence, the potential of prostate cancer (PCa)-derived EVs is being explored as a transformative approach for the management of high-risk prostate cancer.

The project qualifies as a basic research study with potential translational relevance. An observational retrospective study has been designed with the objective of comprehensively characterizing extracellular vesicles (EVs) derived from EPS-urine using multi-omics approaches. The analysis will be conducted on samples from 100 patients, all recruited exclusively at the Department of Urology at IRCCS San Raffaele Hospital. Patients are categorized into two groups: patients with clinically significant prostate cancer (csPCa), including intermediate-risk PCa (ISUP grade 2-3) and high-risk PCa (ISUP grade 4-5), and patients with non-clinically significant PCa (non-csPCa), including low-risk PCa (ISUP grade 1) and patients with benign prostatic hypertrophy. The study is expected to provide unprecedented insights into prostate tissue-derived EVs, laying the foundation for functional validation of key molecular markers and pathways implicated in PCa progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received diagnosis of PCa or BPH through prostate biopsies between 2016 and 2018 and subsequently have signed the informed consent (URBBAN protocol "Regulation for the collection, storage and use of human biological material" v.4 of 14/02/2014 or v.5 of 10/04/2017)
* EPS-urine samples collected from patients undergoing prostate biopsies
* Aged > 18 years old

Exclusion Criteria:

* Aged < 18 years old
* Concomitant other urological malignancies
* Previous systemic oncological treatments for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients who received diagnosis of PCa or BPH through prostate biopsies between 2016 and 2018. EPS-urine samples were collected from all patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Identify a multi-omics signature from EPS-urine derived EVs in prostate cancer | Baseline / Time zero
  The primary objective is to identify a multi-omics signature from EPS-urine derived EVs in prostate cancer. All these analyses will be included:
  1. Multi-Omics characterization of bulk EPS-urine derived EVs
  2. Enrichment for prostate-specific EV subpopulations using specific markers
  3. Optimization of low loads LC-MS/MS methods for analysis of prostate specific EVs
  To achieve the primary objective the following analysis will be performed:
  1. Determination of relative abundance (peak intensities) of EV-associated proteins, lipids and metabolites measured by high-resolution LC-MS/MS
  2. Determination of Purity and concentration (particles/mL) of highly specific prostate derived EVs subpopulation by NTA (nanoparticle tracking analysis) and fluorescence
  3. Determination of relative abundance (peak intensities) and eventual differential pattern of Prostate-specific EVs proteins, lipids and metabolites measured by high-resolution and high throughput mass spectrometer

SECONDARY OUTCOMES:
Correlation between EVs multiomics profiling and prostate cancer clinical progression. | Baseline / Time zero
  The secondary objective is to evaluate if there is a correlation between EVs multiomics profiling and prostate cancer clinical progression.
  To determine this correlation, the patients will be divided in two groups:
  * clinically significant prostate cancer (csPCa), including intermediate-risk PCa (ISUP grade 2-3) and high-risk PCa (ISUP grade 4-5)
  * non-clinically significant PCa (non-csPCa): including low-risk PCs (ISUP grade 1) and patients with benign prostatic hypertrophy.
  Samples will be characterized by multi-comics approaches in LC-MS/MS. The data collected from the two groups will be compared and evaluated using t-test statistical method. Based on the results obtained in this first phase of the study, the next step will be the validation of a predictive model using EVs multi-omics profile and patients' clinical data along with imaging data, through artificial intelligence (AI). This second part will be the object of a future study on an independent cohort of patients.